CLINICAL TRIAL: NCT02314585
Title: Fall Risk Reduction in Multiple Sclerosis: Exercise Intervention vs. Attention Control Modification
Brief Title: Fall Risk Reduction in Multiple Sclerosis (FIRMS)
Acronym: FIRMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 15053
Record Dates: First submitted 2014-11-23; First posted 2014-12-11 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Other): In the second phase, participants will partake in an instructional class relating to gait, balance, and falls.
  Interventions: Other: Education
- Exercise (Other): In the second phase,participants will partake in an exercise course relating to gait, balance, and falls.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will partake in three, six month phases. In the second phase, either an education or exercise program will be implemented. Assessments will follow each phase with the addition of an initial assessment for baseline data.
  Arms: Exercise
Other: Education — Participants will partake in three, six month phases. In the second phase, either an education or exercise program will be implemented. Assessments will follow each phase with the addition of an initial assessment for baseline data.
  Arms: Education

SUMMARY:
This study looks to see the effects of a home based exercise program on falls in people with MS.

DETAILED DESCRIPTION:
The purposes of this project are four-fold: 1) to determine if a 6-month home-based targeted exercise program results in immediate and sustained reduction in falls risk and incidence ; 2) to identify the factors that contribute to a reduction in fall risk and incidence; 3) to determine if a decrease in physiological fall risk and/or fall incidence results in increased quality of life and participation in older adults with MS; and 4) to determine the association between cognition, environment and comorbidities on future falls and intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria involve having an established definite diagnosis of MS
* Ability to walk 25 feet with or without aid
* Relapse free in the last 30 days
* Being ≥ 50 years of age
* Having fallen at least once in the past year
* Physician approval to engage in light physical activity
* Willingness and ability to attend the training sessions and testing sessions.

Exclusion Criteria:

* We will exclude all individuals with risk factors contra-indicative for undertaking strenuous exercise.
* During the initial phone contact with the project coordinator, participants will verbally respond to a health history questionnaire.
* Those individuals who are asymptomatic and meet no more than one risk factor threshold including family history of coronary heart disease, hypertension, high cholesterol, diabetes, obesity, and sedentary lifestyle will be considered at low risk and included for participation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Chagne in Fall Risk | 1 year
  The primary outcome measure of this investigation is physiological fall risk. Physiological fall risk will be determined by the short form of the physiological profile assessment (PPA). The PPA is a validated tool to assess physiological function related to fall risk by combining measures of vision, proprioception, lower-limb strength, postural sway, and cognitive function. It is predictive of future fall risk in persons with MS. The PPA provides a fall risk score that is based on the quantification of key physiological markers (e.g. vision, leg strength, proprioception, balance, cognition, etc) and comparison of those markers to age and gender matched normative data. The PPA provides a therapeutically relevant prognostic predictor of falls and this makes it an ideal outcome measure of investigations evaluating fall prevention strategies.

SECONDARY OUTCOMES:
Identification of Fall Risk Factors | 1 year
  The secondary outcome of fall incidence will be monitored prospectively for 6 months prior to and immediately following the 24 week intervention period via a fall diary A fall will be defined as an event where an individual unintentionally comes to the ground. Participants will receive a biweekly phone call and weekly text to inquire if they have suffered a fall and to remind them to complete the diary. If a fall is reported details of falls, information about injury, and other pertinent information will be attained. The fall diary will be contained in a brightly labeled binder and participants will be asked to mark if they have or have not fallen on a given day. At the end of each month participants will mail the dairy back in a preaddressed prepaid envelope to the research lab. The fall calls/diary will allow for the determination of number of falls, and fall rate per person year.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J Sosnoff, PhD, Principal Investigator — Motor Control Lab, University of Illinois
Locations (1):
- Motor control research lab, Urbana, Illinois, United States